CLINICAL TRIAL: NCT03501979
Title: A Phase II Non-randomized Study to Assess the Safety and Efficacy of the Combination of Tucatinib and Trastuzumab and Capecitabine for Treatment of Leptomeningeal Metastases in HER2 Positive Breast Cancer
Brief Title: Tucatinib, Trastuzumab, and Capecitabine for the Treatment of HER2+ LMD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study accrual ended early due to the FDA approval of tucatinib in metastatic HER2+ breast cancer
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); Johns Hopkins University (Other); Seagen Inc. (Industry); University of Michigan (Other); Georgetown University (Other); University of California, San Francisco (Other); University of Chicago (Other); Indiana University (Other); University of Washington (Other); University of Texas (Other)
Responsible Party: Principal Investigator, Erica Stringer-Reasor, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB 1794
Record Dates: First submitted 2018-04-08; First posted 2018-04-18 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Breast Cancer; Leptomeningeal Disease
Keywords: HER2+; metastatic breast cancer; leptomeningeal disease; tucatinib; trastuzumab; capecitabine
MeSH Terms: conditions — Breast Neoplasms; Meningeal Neoplasms | interventions — tucatinib; Trastuzumab; Capecitabine

STUDY DESIGN:
Intervention Model Description: Subjects will receive combination treatment with tucatinib + trastuzumab + capecitabine every 21 days, which is one cycle. Evaluation will be done every two cycles with an MRI of the brain and spine. Cycles 3 and beyond will be at the discretion of the physician. A scan will be done every four cycles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tucatinib + Trastuzumab + Capecitabine (Experimental): Tucatinib will be taken orally at 300 mg twice a day starting with Cycle 1, Day 1. A cycle consists of 21 days. Capecitabine will be taken orally at 1000 mg/m2 twice a day on Days 1-14 starting with cycle 1. Trastuzumab is given intravenously as a loading dose of 8 mg/kg on Cycle 1, Day 1 and then at 6 mg/kg for all subsequent cycles.
  Interventions: Drug: Tucatinib; Drug: Trastuzumab; Drug: Capecitabine

INTERVENTIONS:
Drug: Tucatinib — Tucatinib study drug is given in tablet form and taken daily.
  Other Names: ONT-380
Drug: Trastuzumab — Trastuzumab is approved by the FDA and is available commercially. Trastuzumab must be prepared and is administered intravenously.
Drug: Capecitabine — Capecitabine is approved by the FDA and is available commercially as an oral drug.

SUMMARY:
A phase 2 non-randomized study to assess the safety and efficacy of the combination of tucatinib and trastuzumab with capecitabine for the treatment of leptomeningeal metastases in HER2-neu positive breast cancer.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a new treatment for patients with HER2+ metastatic breast cancer (MBC) with leptomeningeal disease (LMD). This is a rare and fast-growing form of cancer. Leptomeningeal disease refers to the seeding of tumor cells to the leptomeninges and dissemination in the cerebrospinal fluid.

Currently, there are is no standard of care treatment for LMD. However, we think the combination therapy will be safe and well-tolerated and may also improve survival. Blood and spinal fluid samples will be collected to evaluate the effects on the body and the cancer, which will help provide greater understanding to therapy response in patients.

The study has a two-stage design with the first stage including 15 subjects from up to ten institutions nationwide. If it advances to the second stage based on the number of successes, another 15 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age ≥18 years at time of consent
* Histologically proven metastatic infiltrating carcinoma of the breast that is HER2 positive - Immunohistochemistry (IHC) 3+ and/or Fluorescence in situ hybridization (FISH) ratio >2.0, or average HER2 copy number >6.0 signals per cell or per current ASCO-CAP (American Society of Clinical Oncology - College of American Pathologists) or NCCN (National Comprehensive Cancer Network) guidelines. (NOTE: HER2 testing may be performed on primary and/or metastatic site; Any estrogen and progesterone [ER/PR] status is allowed.)
* Evidence of leptomeningeal disease (LMD) as diagnosed by a) presence of malignant cells in CSF (+CSF cytology) and/or b) Magnetic Resonance Imaging (MRI) evidence of LMD, plus clinical signs and/or symptoms. NOTE: Measurable extra-CNS disease is not required. Note: Patients who have MRI evidence of focal LMD with negative cytology and no symptoms are not eligible for enrollment.
* Karnofsky Performance Status ≥ 50 or Eastern Cooperative Oncology Group (ECOG) ≤ 3
* Patient is able and willing to undergo study-required testing including:

  1. Contrast-enhanced MRI Note: If patient has implants in place that are MRI incompatible, these must be removed prior to enrollment.
  2. Placement of an Ommaya reservoir (ventricular access device). Note: This is mandatory for the first 15 patients enrolled onto the protocol (first stage). In the second stage, this is strongly recommended per protocol. If a patient cannot or chooses not to undergo Ommaya placement in the second stage, the patient will be allowed to enroll.
  3. Evaluation by medical oncologist at baseline and at every cycle (required)
  4. Evaluation by neurologist/neuro-oncologist at baseline and at every cycle (strongly recommended); if this is not possible at a site, a medical oncologist may per perform the protocol specified evaluations at each visit.
* Patients who are on steroids due to CNS disease or LMD diagnosis should be on a stable dose for at least 5 days prior to registration.
* Prior treatment allowances are as follows:

  1. >14 days since last dose of any previous endocrine therapy, chemotherapy, trastuzumab or other antibody-based therapy. NOTE: If patients have been previously receiving trastuzumab on a weekly basis (at a dose of 2mg/kg), only a 7 day washout will be required.
  2. >14 days or five half-lives since previous treatment with any experimental agent, whichever is greater
  3. Cumulative dose of doxorubicin >360 mg/m2 or previous treatment with another anthracycline with cumulative dose equivalent to >360 mg/m2 doxorubicin is not allowed.
  4. Patients must not have received any therapy specifically directed at LMD, including prior systemic or intrathecal therapy for LMD.
  5. Radiotherapy:

     * Patients must not have received radiotherapy to the neuroaxis following diagnosis of LMD for the purpose of treating LMD, and may not receive

       * radiotherapy to the neuroaxis concurrently with the study drug;
     * Patients must not have received whole brain radiotherapy for parenchymal metastases within the last 2 weeks (14 days) or focal CNS radiotherapy within 1 week (7 days) prior to first dose of study drug. Note: Radiation for the purpose of palliation in the setting of a painful bone or dural metastasis can be allowed at the discretion of the treating physicians.
* All toxicity related to prior cancer therapies must have resolved to ≤ Grade 1, with the following exceptions: alopecia; neuropathy, which must have resolved to ≤ Grade 2; and CHF, which must have been ≤ Grade 1 in severity at the time of occurrence, and must have resolved completely. Must be without significant systemic illness (e.g. infection unresponsive to treatment after 7 days)
* Adequate hematologic, liver, and renal function, as follows:

  1. Hemoglobin ≥ 9 g/dL
  2. ANC ≥ 1000 cells/μL
  3. Platelets ≥ 100,000/μ
  4. Total bilirubin ≤ 1.5 X upper limit of normal (ULN), unless a known history of Gilbert's disease (≤ 3 X ULN)
  5. Transaminases (AST/SGOT and ALT/SGPT) ≤ 2.5X ULN (< 5 X ULN if liver metastases are present)
  6. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 X ULN
  7. Creatinine clearance (CrCL) ≥ 50 mL/min
* Left ventricular ejection fraction (LVEF) must be within institutional limits of normal as assessed by ECHO or MUGA documented within 4 weeks prior to enrollment on the study.
* Able to understand the study requirements and document informed consent indicating his/her awareness of the investigational nature and the risks of this study.

Exclusion Criteria:

* Medical, social, or psychosocial factors that, in the opinion of the Investigator, could impact safety or compliance with study procedures.
* Patient is pregnant or is breastfeeding. Note: If female and of child-bearing potential (females who are not surgically sterile or who have had a period in the last 12 months), has negative pregnancy test within 21 days prior to treatment. If a sexually active male or a sexually active female of child- bearing potential, agrees to use dual (two concurrent) forms of medically accepted contraception from the time of consent until 6 months after the last dose.
* History of allergic reactions to compounds of similar chemical or biological composition to capecitabine (Group A only), trastuzumab or tucatinib, except for a history of Grade 1 or Grade 2 infusion related reaction to trastuzumab, that has been successfully managed.
* Known to be HIV positive, or a carrier for Hepatitis B and/or Hepatitis C (whether active disease or not)
* Known liver disease, autoimmune hepatitis, or sclerosing cholangitis
* Inability to swallow pills or any significant gastrointestinal diseases, which would preclude adequate absorption of oral medications
* Use of a strong CYP2C8/CYP3A4 inducer or inhibitor within three elimination half-lives of the inducer or inhibitor prior to the start of study treatment.
* Known impaired cardiac function or clinically significant cardiac disease such as ventricular arrhythmia requiring therapy or congestive heart failure. Note: Patients with hypertension must have controlled disease defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg on antihypertensive medications.
* Myocardial infarction or unstable angina within 6 months prior to the first dose of study drug.
* Patient with known dihydropyrimidine dehydrogenase deficiency
* Previous treatment with tucatinib
* Previous treatment with capecitabine within 12 months prior to study registration
* Prior history of other cancer (except non melanoma skin, cervical intraepithelial neoplasia) with evidence of disease within the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica M Stringer-Reasor, MD, Principal Investigator — University of Alabama at Birmingham; Rashmi K Murthy, MD, MBE, Study Chair — M.D. Anderson Cancer Center; Barbara J O'Brien, MD, Study Chair — M.D. Anderson Cancer Center
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCSF-Mission Bay, San Francisco, California
  - MedStar Georgetown University-Lombardi CCC, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Indiana University-Melvin and Bren Simon cancer center, Indianapolis, Indiana
  - Dana Farber/Harvard Cancer Center-, Boston, Massachusetts
  - University of Michigan-, Ann Arbor, Michigan
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center-Montlake, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tucatinib + Trastuzumab + Capecitabine
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tucatinib + Trastuzumab + Capecitabine
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 53 [33 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17
Patient Demographics [Count of Participants; unit: Participants] | 17

OUTCOME MEASURES:

1. Primary Outcome: Length of Subject Survival After Starting Study Treatment
Description: Number of participants alive. A Gehan-like trial design with an interim futility analysis will be used.
Time Frame: Through study completions, an average of 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Tucatinib + Trastuzumab + Capecitabine
Number analyzed (Participants) | 17
Participants | 6

2. Secondary Outcome: Number of Adverse Events
Description: Adverse event reporting will be graded following the National Cancer Institute of Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0. Subjects who receive at least one dose of the drug combination will be evaluable for toxicity from the time of the first dose.
Time Frame: up to 28 months
Measure: Number; unit: participants
Arm/Group | Tucatinib + Trastuzumab + Capecitabine
Number analyzed (Participants) | 17
participants
  diarrhea | 13
  fatigue | 9
  nausea/vomiting | 8
  hand-foot syndrome | 13
  liver function test elevation | 11

3. Secondary Outcome: Progression Free Survival
Description: From the start of treatment to 12 months
Time Frame: up to 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tucatinib + Trastuzumab + Capecitabine
Number analyzed (Participants) | 17
months | 10 [4.1 to 10]

4. Secondary Outcome: Duration of Response in the Central Nervous System (CNS)
Description: Data from subjects who have received at least one cycle of therapy and disease re-evaluation for CNS tumors by imaging, cytopathology, and clinical evaluation will be accumulated until disease progression.
Time Frame: up to 28 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tucatinib + Trastuzumab + Capecitabine
Number analyzed (Participants) | 17
months | 6.9 [2.8 to 13.8]

5. Secondary Outcome: Clinical Benefit Rate (CBR) in CNS
Description: The overall survival from the combination therapy is compared to the historical control. Clinical benefit is observed with a ratio of successes and corresponding confidence interval.
Time Frame: Baseline up to 28 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tucatinib + Trastuzumab + Capecitabine
Number analyzed (Participants) | 17
Participants | 6

6. Secondary Outcome: Duration of Response in Extra-CNS Disease
Description: Data from subjects who have received at least one cycle of therapy and disease re-evaluation for extra-CNS tumors by imaging, cytopathology, and clinical evaluation will be accumulated until disease progression. Extra-CNS response will be classified per the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: up to 28 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tucatinib + Trastuzumab + Capecitabine
Number analyzed (Participants) | 17
months | 4.1 [2.3 to 11.4]

7. Secondary Outcome: Clinical Benefit Rate (CBR) in Extra-CNS Disease
Description: as for outcome 5
Time Frame: up to 28 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tucatinib + Trastuzumab + Capecitabine
Number analyzed (Participants) | 17
Participants | 6

8. Secondary Outcome: Symptom Burden
Description: The M.D. Anderson Symptom Inventory Brain Tumor (MDASI -BT) module questionnaire will collect data at each study time point and evaluate changes of symptom burden. The MDASI-BT scale measures the severity of symptoms experienced by patients with breast cancer that interfere with daily living. A greater number of symptoms equals a greater interference with daily living. Symptoms of severity are assessed on a 0-213 scale with 0 being "lower quality of life" and 213 "higher quality of life".
Time Frame: Baseline, end of study (up to 28 months)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tucatinib + Trastuzumab + Capecitabine
Number analyzed (Participants) | 12
score on a scale
  baseline | 61 [0 to 213]
  end of study | 32 [0 to 213]

9. Secondary Outcome: Quality of Life Assessment
Description: The Linear Analog Scale Assessment Quality of Life will be used to evaluate changes in the quality of life at restaging visits.
  Scale ranges from 0 to 100. Higher scores indicate a better quality of life.
Time Frame: up to 28 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tucatinib + Trastuzumab + Capecitabine
Number analyzed (Participants) | 17
score on a scale | 31 [11 to 47]

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events while on study drugs and up to 1 month after discontinuation of study drug (up to 28 months).
Arm/Group | Tucatinib + Trastuzumab + Capecitabine
All-Cause Mortality (participants affected / at risk) | 11/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tucatinib + Trastuzumab + Capecitabine (N=17)
Elevated liver function test (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tucatinib + Trastuzumab + Capecitabine (N=17)
Diarrhea (Gastrointestinal disorders) | 13 (13)
Fatigue (General disorders) | 10 (10)
Nausea/Vomiting (Gastrointestinal disorders) | 10 (10)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 13 (13)
Elevated liver function test (Gastrointestinal disorders) | 11 (11)

LIMITATIONS AND CAVEATS:
The study only remains open to monitor patients for overall survival per the primary endpoint after FDA approval was granted for tucatinib in advanced stage HER2+ breast cancer in April 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03501979/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03501979/ICF_001.pdf